CLINICAL TRIAL: NCT03863743
Title: Impact of Integrated Care Pathways for Prevention of Post-operative Urinary Retention in Primary Total Knee or Total Hip Replacement: Prospective Randomized Control Trial
Brief Title: Impact of Integrated Care Pathways for Prevention of Post-operative Urinary Retention (POUR)
Acronym: POUR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TriHealth Inc. (Other)
Responsible Party: Principal Investigator, Mark Snyder, Principal Investigator, TriHealth Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-012
Record Dates: First submitted 2019-03-03; First posted 2019-03-05 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee; Urinary Retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Intervention Model Description: 164 patients will be randomized to either the control group or the experimental group. Patients will be randomized immediately following the signed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Patient will complete IPSS score, medical history, and risk factors for POUR will be evaluated. Patient will undergo treating physician's standard of care for total hip or knee replacement. Patient will receive bladder scans in PACU, upon admission to the nursing unit, and prior to discharge (post-void).
  Interventions: Other: physician's standard of care
- Experimental (Experimental): Patient will complete IPSS score, medical history, and risk factors for POUR will be evaluated. If considered high risk (determined by IPSS), then patient Patient will undergo integrated care pathway that avoids narcotics. Bladder volume will be measured in PACU, after admission to the nursing unit, and prior to discharge from the hospital (post-void).
  Interventions: Other: integrated care pathway

INTERVENTIONS:
Other: integrated care pathway — Incidence of POUR after undergoing total hip or knee replacement and integrated care pathway will be evaluated.
  Arms: Experimental
Other: physician's standard of care — Incidence of POUR will be evaluated in standard of care treatment.
  Arms: Control

SUMMARY:
A prospective randomized control trial will be conducted at Good Samaritan Hospital and TriHealth Evendale Hospital. Subjects will receive total hip or knee surgery and follow-up via standard care at the discretion of the treating physician or the experimental study arm in which all patients will undergo the integrated care pathway.

DETAILED DESCRIPTION:
Patients will be randomized to the control group or the experimental group. Patients in the control group will receive the treating physician's standard of care, and undergo bladder scans in the post anesthesia care unit (PACU), upon admission to the unit, and prior to discharge from the hospital. Patients in the experimental group will undergo a multimodal pain control care pathway that minimizes opioid consumption.

The primary endpoint will be the presence of or absence of post-operative urinary retention (POUR) between discharge from the PACU and prior to discharge from the hospital. POUR will be defined as bladder volume of greater than 500cc and the inability to void for at least 2 hours within the first 24 hours. POUR, once identified will be treated with intermittent straight catheterization (ISC). Secondary endpoints will include opioid consumption (in morphine milligram equivalents; MME), genito-urinary consultation, type (knee or hip) and duration of surgery, type of anesthesia, duration of anesthesia, total amount of IV fluids, blood loss, length of hospital stay (LOS), discharge status (home with early outpatient physical therapy, etc.), time of first spontaneous voiding, and the number of ISCs and any necessary indwelling catheterization and adverse events of interest including POUR, post-operative nausea and vomiting (PONV), severe pain of 7 or greater on the numeric rating scale(NRS), blood loss requiring transfusion, and lower urinary tract symptoms (LUTS).

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I- III
* BMI under 36 kg/m^2
* Scheduled surgery for primary total hip or knee replacement
* Age 18+ years

Exclusion Criteria:

* Contraindications or failure of neuraxial anesthesia
* Patients must not be outpatient total hip or knee procedure
* Known intercurrent UTI, incontinence, or urinary retention not addressed by pre-operative urologic consultation and correction
* Pregnancy
* Current nicotine, alcohol or drug abusers
* Pre-operative narcotic use (any narcotic consumption within 3 days prior to surgery)
* Post- operative parenteral narcotic administration
* Allergy or intolerance to liposomal bupivacaine, bupivacaine, celecoxib, dexamethasone and/or pregabalin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2022-02-05 (Estimated); Study Completion 2022-02-05 (Estimated)

PRIMARY OUTCOMES:
POUR | up to 24 hours post-op
  presence or absence of urinary retention

SECONDARY OUTCOMES:
opioid consumption | up to 14 days following the joint procedure
  opioid consumption (in morphine milligram equivalents; MME)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Snyder, MD, Principal Investigator — TriHealth Inc.
Locations (2):
- United States (2):
  - TriHealth Good Samaritan Hospital, Cincinnati, Ohio
  - TriHealth Evendale Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No
IDP will not be available to other researchers

REFERENCES:
- [Background] Hollman F, Wolterbeek N, Veen R. Risk Factors for Postoperative Urinary Retention in Men Undergoing Total Hip Arthroplasty. Orthopedics. 2015 Jun;38(6):e507-11. doi: 10.3928/01477447-20150603-59. PMID 26091224
- [Background] Umer A, Ross-Richardson C, Ellner S. Incidence and Risk Factors for Postoperative Urinary Retention: A Retrospective, Observational Study with a Literature Review of Preventive Strategies. Conn Med. 2015 Nov-Dec;79(10):587-92. PMID 26731878
- [Background] Baldini G, Bagry H, Aprikian A, Carli F. Postoperative urinary retention: anesthetic and perioperative considerations. Anesthesiology. 2009 May;110(5):1139-57. doi: 10.1097/ALN.0b013e31819f7aea. PMID 19352147
- [Background] Cronin JJ, Shannon FJ, Bale E, Quinlan W. Prediction of post-operative urinary retention in hip and knee arthroplasty in a male population. European Journal of Orthopaedic Surgery & Traumatology. 2007;17(1):47-50.
- [Background] Fazeli F, Gooran S, Taghvaei ME, Fazeli K. Evaluating International Prostate Symptom Score (IPSS) in Accuracy for Predicting Post-Operative Urinary Retention After Elective Cataract Surgery: A Prospective Study. Glob J Health Sci. 2015 Mar 26;7(7 Spec No):93-6. doi: 10.5539/gjhs.v7n7p93. PMID 26153208
- [Background] Akkoc A, Aydin C, Topaktas R, Kartalmis M, Altin S, Isen K, Metin A. Prophylactic effects of alpha-blockers, Tamsulosin and Alfuzosin, on postoperative urinary retention in male patients undergoing urologic surgery under spinal anaesthesia. Int Braz J Urol. 2016 May-Jun;42(3):578-84. doi: 10.1590/S1677-5538.IBJU.2015.0256. PMID 27286124
- [Background] Brouwer TA, Eindhoven BG, Epema AH, Henning RH. Validation of an ultrasound scanner for determing urinary volumes in surgical patients and volunteers. J Clin Monit Comput. 1999 Aug;15(6):379-85. doi: 10.1023/a:1009939530626. PMID 12578033
- [Background] Tischler EH, Restrepo C, Oh J, Matthews CN, Chen AF, Parvizi J. Urinary Retention is Rare After Total Joint Arthroplasty When Using Opioid-Free Regional Anesthesia. J Arthroplasty. 2016 Feb;31(2):480-3. doi: 10.1016/j.arth.2015.09.007. Epub 2015 Sep 18. PMID 26453530
- [Background] Gerrard AD, Brooks B, Asaad P, Hajibandeh S, Hajibandeh S. Meta-analysis of epidural analgesia versus peripheral nerve blockade after total knee joint replacement. Eur J Orthop Surg Traumatol. 2017 Jan;27(1):61-72. doi: 10.1007/s00590-016-1846-z. Epub 2016 Sep 3. PMID 27592218
- [Background] Dysart S, Snyder MA, Mont MA. A Randomized, Multicenter, Double-Blind Study of Local Infiltration Analgesia with Liposomal Bupivacaine for Postsurgical Pain Following Total Knee Arthroplasty: Rationale and Design of the Pillar Trial. Surg Technol Int. 2016 Nov 11;30:261-267. PMID 27824434
- [Background] Mont MA, Beaver WB, Dysart SH, Barrington JW, Del Gaizo DJ. Local Infiltration Analgesia With Liposomal Bupivacaine Improves Pain Scores and Reduces Opioid Use After Total Knee Arthroplasty: Results of a Randomized Controlled Trial. J Arthroplasty. 2018 Jan;33(1):90-96. doi: 10.1016/j.arth.2017.07.024. Epub 2017 Jul 25. PMID 28802777
- [Background] Backes JR, Bentley JC, Politi JR, Chambers BT. Dexamethasone reduces length of hospitalization and improves postoperative pain and nausea after total joint arthroplasty: a prospective, randomized controlled trial. J Arthroplasty. 2013 Sep;28(8 Suppl):11-7. doi: 10.1016/j.arth.2013.05.041. Epub 2013 Aug 9. PMID 23937923
- [Background] Snyder MA, Scheuerman CM, Gregg JL, Ruhnke CJ, Eten K. Improving total knee arthroplasty perioperative pain management using a periarticular injection with bupivacaine liposomal suspension. Arthroplast Today. 2016 Jan 11;2(1):37-42. doi: 10.1016/j.artd.2015.05.005. eCollection 2016 Mar. PMID 28326395
- [Background] Boonstra AM, Stewart RE, Koke AJ, Oosterwijk RF, Swaan JL, Schreurs KM, Schiphorst Preuper HR. Cut-Off Points for Mild, Moderate, and Severe Pain on the Numeric Rating Scale for Pain in Patients with Chronic Musculoskeletal Pain: Variability and Influence of Sex and Catastrophizing. Front Psychol. 2016 Sep 30;7:1466. doi: 10.3389/fpsyg.2016.01466. eCollection 2016. PMID 27746750
- [Background] Balderi T, Carli F. Urinary retention after total hip and knee arthroplasty. Minerva Anestesiol. 2010 Feb;76(2):120-30. PMID 20150853
- [Background] Maheshwari AV, Boutary M, Yun AG, Sirianni LE, Dorr LD. Multimodal analgesia without routine parenteral narcotics for total hip arthroplasty. Clin Orthop Relat Res. 2006 Dec;453:231-8. doi: 10.1097/01.blo.0000246545.72445.c4. PMID 17031312